CLINICAL TRIAL: NCT00312832
Title: A Randomized Open Label Study Comparing the Impact of Reducing the Dose of Stavudine Versus Switching to Tenofovir on Plasma Lipids, Body Composition and Mitochondrial Function in HIV-Infected Patients Receiving Antiretroviral Therapy
Brief Title: Study Comparing Reducing the Dose of Stavudine Versus Switching to Tenofovir in HIV-Infected Patients Receiving Antiretroviral Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D40-30
Record Dates: First submitted 2006-04-07; First posted 2006-04-11 (Estimated); Last update posted 2006-10-24 (Estimated); Status verified 2004-01

CONDITIONS: HIV Infections; Lipoatrophy
Keywords: HIV; d4T; TDF; lipoatrophy; treatment experienced; HIV-infection
MeSH Terms: conditions — HIV Infections; Lipodystrophy; Acquired Immunodeficiency Syndrome | interventions — Drug Tapering

INTERVENTIONS:
Drug: switching; dose reduction

SUMMARY:
Background: Stavudine-containing regimens are associated with a potential for lipoatrophy and dyslipidemia. We assessed the safety and efficacy of reducing the dose of stavudine compared to switching to tenofovir or maintaining the standard dose of stavudine.

Methods: Clinically stable lipoatrophic HIV-infected patients receiving antiretroviral therapy containing stavudine 40 mg bid with a plasma HIV RNA <200 copies/mL for at least 6 months were randomized to maintain stavudine 40 mg bid (d4T40 arm), to reduce to 30 mg bid (d4T30 arm), or to switch from stavudine to tenofovir-DF (TDF arm) while preserving the remaining drugs. Fasting metabolic parameters were assessed at baseline and at weeks 4, 12, and 24. Mitochondrial parameters in peripheral blood mononuclear cells and body composition were measured at baseline and at week 24.

ELIGIBILITY:
Inclusion Criteria:

Study eligibility criteria included documented HIV infection, age 18 years or older, moderate to severe clinical lipoatrophy in at least one region upon physical examination (17,18), viral load <200 copies/mL for at least 6 months prior to inclusion in the study, and a stable triple antiretroviral therapy including d4T 40 mg bid for at least the 6 preceding months, and no prior TDF use.

Exclusion Criteria:

Prior TDF use, viral load>200 copies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-01; Study Completion 2005-02

CONTACTS AND LOCATIONS:
Overall Officials: Jose Maria Gatell, Principal Investigator — Hospital Clinic of Barcelona